CLINICAL TRIAL: NCT05541640
Title: Effect of Intraoperative Lidocaine Infusion on Inducing Intestinal Motility and Surgery-induced Release of Pro-inflammatory Cytokines After Abdominal Surgery. A Prospective, Comparative, Randomized Double Blind Controlled Clinical Study
Brief Title: Intraoperative Lidocaine Infusion and Surgery-induced Release of Pro-inflammatory Cytokines After Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, asisstant lecturer of anaesthesia and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: zzzz
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator)
  Interventions: Drug: normal saline group
- lidocaine group (Active Comparator)
  Interventions: Drug: lidocaine group

INTERVENTIONS:
Drug: normal saline group — normal saline infusion at the start of surgery
  Arms: control group
Drug: lidocaine group — lidocaine infusion at the start of surgery
  Arms: lidocaine group

SUMMARY:
Lidocaine is an amide local anaesthetic and an antiarrhythmic agent, first synthesized in 1942, and after approval for human use was launched in 1948 in Sweden The first observations of post operative analgesic effects of perioperative intravenous lidocaine (IVL) were initially proposed in 1951 subsequently many more enthusiastic reports followed. Postoperative formal clinical evaluations in the perioperative setting were conducted in the late 1950s where IV Lidocaine was demonstrated to have a postoperative analgesic effect without posing the risk of respiratory depression, reducing the occurrence of postoperative nausea and vomiting (PONV), and enhance post-surgical recovery. IV Lidocaine also potentiated the depth of anesthesia and led to a better tolerance of endotracheal intubation.Around 40% of patients experience a delay in resumption of normal bowel function after colorectal surgery. This delay leads to symptoms of nausea, vomiting, constipation, and abdominal distension, which then require unpleasant supportive interventions such as intravenous fluids and nasogastric tube insertion. There is no remedy to address this delay. ALLEGRO, "A placebo-controlled randomized trial of intravenous Lidocainein accelerating Gastrointestinal Recovery surgery," is the latest ongoing multicenter research study across the United Kingdom, investigating the use of intravenous lidocaine to improve recovery after colorectal surgery

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Both sexes, males and females
* Patients scheduled for elective intestinal surgery.
* Body mass index (BMI) 18-30 kg•m-2.
* ASA I - II.

Exclusion Criteria:

* Patient refusal
* Patients with preoperative gastrointestinal dysfunction.
* Patients with a history of drug abuse, or long-term opioid use.
* ASA III and VI
* Patients with a history of previous gastrointestinal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
postoperative visual analogue score (VAS SCORE) | 24 hour
  assessment of postoperative pain will be carried by VAS in which zero=no pain and 10= worst pain ever

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt